CLINICAL TRIAL: NCT04218305
Title: Study of Using Serum Fetuin-A as a Marker in Obesity and Type 2 Diabetes Mellitus
Brief Title: Fetuin-A as a Marker in Obesity and Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosam Mohammad Ahmad, Dr., Minia University
Other Study IDs: fetuin-A as a marker
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- The first group: Include One hundred patients with type 2 diabetes mellitus with average body mass index.
  Interventions: Diagnostic Test: Serum Level Of Fetuin A
- The second group: Include One hundred patients whose body mass index is 30 or over without diabetes.
  Interventions: Diagnostic Test: Serum Level Of Fetuin A
- The third group: Include One hundred type 2 diabetic obese patients whose body mass index is 30 or over.
  Interventions: Diagnostic Test: Serum Level Of Fetuin A
- The fourth group: Include One hundred apparently healthy adult person as a control.
  Interventions: Diagnostic Test: Serum Level Of Fetuin A

INTERVENTIONS:
Diagnostic Test: Serum Level Of Fetuin A

SUMMARY:
The aim of this study is to assess the significance of serum fetuin-A as a marker of obesity and type 2 diabetes mellitus. We used multiple statistical approaches to determine that the fetuin-A level is correlated to body mass index (BMI) as well as random blood sugar in type 2 diabetic patients. Also, we found that there is a Positive correlation between the serum fetuin-A levels and the level of glycosylated hemoglobin (HbA1c) in diabetic patients.

DETAILED DESCRIPTION:
The study was a case-control study. We started the study to be performed on eighty subjects divided into four groups:

The first group: include twenty subjects with type 2 diabetes mellitus The second group: include twenty obese subjects whose body mass index is 30 or over The third group: include twenty obese subjects with type 2 diabetes mellitus The fourth group includes twenty apparently healthy subjects as control.

In this study, we concluded that:

1. Serum fetuin-A can be used as a biomarker and independent risk factor and marker for diagnosis of DM and DM has a detrimental effect on serum fetuin-A fetuin-A could be of relevance for the development of insulin resistance
2. Higher fetuin-A concentrations were associated with type 2 diabetes and insulin resistance
3. Increased serum fetuin-A levels constitute an independent marker of lipid profile.
4. fetuin-A may play a role in the pathogenesis of T2DM.
5. The inhibition of insulin receptor by fetuin-A may lead to increased lipolysis and efflux of free fatty acids from adipose tissue. This could explain associated dyslipidemia observed in type 2 diabetic patients in the present study.

Finally, our finding that high plasma fetuin-A levels predict the incidence of type 2 diabetes independently of other established risk factors supports the hypothesis that fetuin-A may play a role in the development of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* • The study included obese and type 2 diabetic patients aged 45-60 years old. and control healthy adult persons

Exclusion Criteria:

* • Cardiac disease and Hypertensive disease

  * Respiratory disease
  * Renal disease
  * GIT and Liver disease
  * Rheumatologic disease
  * Blood disease
  * Endocrine disease except for type 2 diabetes mellitus
  * All with a specific therapeutic drug history.

Ages: 45 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: obese and type 2 diabetic patients aged 45-60 years old. and control healthy adult persons
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
1- Study of human serum fetuin-A and whether it is involved in insulin resistance | Baesline
  2- To assess the significance of serum fetuin-A as a marker in obesity and type 2 diabetes mellitus